CLINICAL TRIAL: NCT05471479
Title: CHARPP (Activated CHARcoal in Poisoned Patient): RCT Pilot Study
Brief Title: Activated CHARcoal in Poisoned Patient - Pilot Trial
Acronym: CHARPP-Pilot
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); VITAM - Centre de recherche en santé durable (Unknown); CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Maude St-Onge, Associate Professor, Clinician-scientist, Laval University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CHARPP - pilot study
Record Dates: First submitted 2022-07-14; First posted 2022-07-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-03

CONDITIONS: Charcoal, Decontamination, Poisoning
Keywords: activated charcoal; decontamination; poisoning; intoxication; toxicity; clinical trial; toxicology; Emergency medicine; PROBE trial
MeSH Terms: conditions — Anthrax; Poisoning | interventions — Charcoal

STUDY DESIGN:
Intervention Model Description: The CHARPP pilot trial employs a Prospective Randomized Open Blinded End-point (PROBE) interventional study model. The study is designed to follow participants forward in time after their enrollment, with interventions and outcomes measured as they occur. Participants are randomly assigned to either the intervention group, which receives activated charcoal, or the control group, which does not receive activated charcoal. This randomization helps to minimize selection bias and balance known and unknown confounding factors across the study groups. The nature of the intervention (activated charcoal) makes it impractical to blind the participants or the clinicians administering the treatment, as the substance visibly changes the color of the oral mucosa to black. While the immediate caregivers and participants know the treatment allocation due to the visible nature of activated charcoal, the outcome assessors and data analysts are blinded to the group assignment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data Analysts: These individuals are responsible for processing and analyzing the collected data. They are blinded to the group allocations to ensure that their analyses are unbiased.
  Research Assistants: Those involved in collecting trial data from participants, including demographics, medical history, and treatment outcomes, are also blinded to the allocation groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AC administration (Experimental): Participants will receive 1g/kg up to a maximum of 50g of activated charcoal by mouth or by naso-gastric tube. The intervention is giving over 15 minutes, as recommended. Activated charcoal can be mixed in a black soft drink to improve palatability and treatment adherence which is often done in usual practice.
  Interventions: Drug: Activated Charcoal
- No AC (Active Comparator): Participants will not receive any activated charcoal
  Interventions: Other: No activated charcoal

INTERVENTIONS:
Drug: Activated Charcoal — Activated charcoal
  Other Names: AC
  Arms: AC administration
Other: No activated charcoal — No activated charcoal
  Arms: No AC

SUMMARY:
The goal of this clinical pilot trial is to determine the feasibility of the clinical trial. Then the large-scale CHARPP will be conducted in order to determine the efficacity of activated charcoal as a treatment for acute poisoning in a diverse population of both adults and children suspected of ingesting toxic substances that activated charcoal can adsorb. The main questions it aims to answer are:

* Can activated charcoal administered within a specific time frame prevent the progression of toxicity?
* How does activated charcoal affect the length of stay in the hospital and the intensive care unit? Researchers will compare the intervention arm (receiving activated charcoal) to the control arm (receiving standard supportive care) to see if activated charcoal reduces hospital stay duration, ICU stay and improves overall patient outcomes.

Participants will:

* Be randomly assigned to either receive activated charcoal or standard supportive care.
* Undergo assessments using standardized clinical scales such as the Poison Severity Score and, for children, the PELODS score.
* Have their functional outcomes evaluated, such as the ability to return to their original residence without help and manage personal hygiene tasks independently.

This structured approach will help clarify the role of activated charcoal in clinical toxicology and inform future treatment protocols.

DETAILED DESCRIPTION:
BACKGROUND: Activated charcoal (AC) is one of the interventions more frequently recommended by poison centers. For instance, in 2020, 32,646 poisoned patients were treated with AC in the United States. This decontamination method has the potential to prevent toxicity and to decrease its severity, but its use is also associated with adverse effects and has a poor palatability. Therefore, we developed a research program named CHARPP (activated CHARcoal in Poisoned Patients) aiming to describe the effect and potential risks associated with the use of AC. This study is particularly focused on whether early administration of activated charcoal can reduce the severity of poisoning outcomes, shorten hospital stays, and mitigate healthcare costs.The first phase of our research program included: a retrospective study and a validation of the Poison Severity Score. The last phase includes a randomized controlled trial (RCT) preceded by a feasibility study in adults and children to compare outcomes in patients who received AC vs those who did not.

OBJECTIVES: This concerns the CHARPP RCT feasibility study which aims to evaluate the possibility of conducting a large multicenter RCT comparing outcomes between poisoned patients who received AC and who did not received AC. The targeted primary outcomes includes: 1) recruitment success (100 patients total at the poison centre associated with hospitals and greater than one patient enrolled/hospital/month), 2) protocol adherence (at least 85% of the patient randomized in the intervention group received AC in less than two hours after group allocation if AC was recommended or did not received it if it was not recommended) and, 3) Less than 5% loss to follow-up. As for the large-scale clinical trial if pilot trial shows feasability, the primary outcome will be progression of toxicity as measured using the Poison Severity Score, a patient-oriented metric frequently used in toxicology; mortality, length of stay in both the intensive care unit and hospital, quality of life as measured by the EQ-5D-5L, and changes in the SOFA score for adults and the PELODS score for children.

METHODS: This randomized concealed multicenter trial will take place in one poison centre and five academic hospitals within the provincial network of the centre antipoison du Québec. Patients presenting to the Emergency rooms with a proven or suspected ingestion of a substance absorbed by activated charcoal and the ones who can receive the intervention within 6 hours of proven or suspected intoxication will be included. Patients requiring or who will likely require another gastro-intestinal decontamination method, who have a contraindication to receive AC, or who ingested a substance with an entero-hepatic circulation requiring multi-dose AC will be excluded. Once the poison centre has identified an eligible patient, we will use a web-based system to perform a randomization in random blocks of two or four. Co-interventions will be standardized as per the poison centre protocols. Follow up will be done every 8h by the poison centres who will also collect data regarding progression of toxicity and relevant outcomes. The research assistant who will extract data will be blinded to study allocation. Only a descriptive analysis will be done for the pilot trial. Data from paediatric patients will be analysed separately. A data and safety monitoring board independent from the study group will follow the results and approve or not the continuation of the study.

RELEVANCE: This will be an excellent opportunity to develop collaborations between poison centers and key actors who will be involved in a larger trial. The results of the research program CHARPP have the potential to influence policies, poison centers recommendations, clinicians' practices and to improve poisoned patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients who presented to the hospital less than 6h after the ingestion of a potentially toxic dose of a carbo-adsorbable substance (substance adsorbed by activated charcoal ).
* Patients who can receive the intervention within 6 hours of proven or suspected intoxication

Exclusion Criteria:

* Patients requiring or who will likely require another gastro-intestinal decontamination method;
* Patients who have contraindication to the use of activated charcoal;
* Patients who ingested a substance with an entero-hepatic circulation requiring multi-dose AC;
* Patients who have no clinical equipoise for the use of activated charcoal as per the attending physician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment success | 12 months
  100 patients total at the poison centre associated with hospitals and greater than one patient enrolled/hospital/month
Protocol adherence | 12 months
  at least 85% of the patient randomized in the intervention group
lost to follow-up | 12 months
  less than 5%

SECONDARY OUTCOMES:
Progression of toxicity (descriptive measure of delta Poison Severity Score - PSS max - PSS at randomization calculated at the end of each case) | 3 months
  measured by the delta Poison Severity Score (min = 0 - better outcome; max = 4 - worse outcome) (and the SOFA - sequential organ failure assessment - score for adults or PELOD -paediatric logistic organ dysfunction - score for children) and available drug levels
Mortality | 3 months
  Will be documented by both the poison centre and the hospitals. Will be collected in by the research coordinator
Length of stay in the intensive care unit and hospital | 3 months
  Will be documented by both the poison centre and the hospitals. Will be collected in by the research coordinator
Duration of mechanical ventilation | 3 months
  Will be documented by both the poison centre and the hospitals. Will be collected in by the research coordinator
functional outcomes (descriptive measure: "back to baseline" or "not back to baseline" calculated at the moment of medical discharge, death or decision of withdrawal of life support) | 6 months
  The ability of patients to return to their daily lives and activities after treatment. Specifically, the trial looks at whether patients can return to their original residence without help and manage personal hygiene tasks such as toileting independently. Will be documented by both the poison centre and the hospitals. Will be collected in by the research coordinator
adverse events | 3 months
  Will be documented by both the poison centre and the hospitals. Will be collected in by the research coordinator

CONTACTS AND LOCATIONS:
Overall Officials: Maude St-Onge, MD PhD FRCPC, Principal Investigator — CHU de Québec - Université Laval
Locations (1):
- CHU de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Feb 2025 up to 6months after publication
Access Criteria: Any scientists